

## STATISTICAL ANALYSIS PLAN

The results of bar overdentures BOD and ball joint overdenture BJOD will be compare for the determination of Ra and the adherence of mold and yeast and mesophyll aerobe. For this, will be used the statistics Shapiro-Wilk, T and the Pearson Correlation Coefficient to determinate the relationship between the study variables. For data processing and analysis the Software Package for Social Sciences (SPSS) version 24.0 will be used.